CLINICAL TRIAL: NCT05350059
Title: Study of High Intensity Focused Ultrasound (HIFU) in the Treatment of Early Breast Cancer
Brief Title: The HIFUB Study (HIFU in Breast Cancer)
Acronym: HIFUB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 233756
Record Dates: First submitted 2022-03-01; First posted 2022-04-27 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Breast Cancer
Keywords: breast cancer; high intensity frequency ultrasound
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: High Intensity Focused Ultrasound (HIFU) treatment to breast cancer
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High Intensity Focused Ultrasound (HIFU) treatment to breast cancer (Experimental): High-Intensity Focused Ultrasound (HIFU) in the Treatment of Early Breast Cancer prior to surgical resection
  Interventions: Device: High Intensity Focused Ultrasound (HIFU) to the Breast Cancer

INTERVENTIONS:
Device: High Intensity Focused Ultrasound (HIFU) to the Breast Cancer — Breast cancer will be ablated using high intensity frequency ultrasound prior to breast surgery

SUMMARY:
High Intensity Focused Ultrasound (HIFU) is a new method of treating solid tumours by thermally ablating them. It has been used in a number of different types of cancers but there is little information on its use in invasive breast cancer (IBC). The investigators aim to assess the efficacy and safety of HIFU in the treatment of IBC.

In this study, fifteen otherwise healthy women diagnosed with small, early stage IBC will be treated with HIFU prior to conventional surgical treatment. The effects of HIFU on the resected tumour will be analysed pathologically and correlated with radiological findings. Immune response and participant experience will also be evaluated

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the trial.
* Female, aged 18 years or above.
* Histologically confirmed breast cancer (invasive ductal cancer) by core biopsy, which is suitable for surgical resection.
* Participants must have one non-metastatic, clinically palpable, invasive breast cancer measuring ≤2cm in its largest dimension, which can be visualised using diagnostic ultrasound.
* All participants must have an adequate biopsy determination of oestrogen, progesterone, HER2 receptor status on pre-operative biopsy.
* Adequate ECG, haematological, renal and hepatic function, as indicated, as would be required for imaging and surgery.
* In the Investigator's opinion, is able and willing to comply with all trial requirements.

Exclusion Criteria:

* Female participant who is pregnant.
* Significant renal or hepatic impairment.
* An inadequate biopsy determination of oestrogen, progesterone, HER2 receptor status on pre-operative biopsy.
* Unable to visualize lesion or tumour boundaries clearly on ultrasound.
* Subjects with tumours lying less than 5mm to overlying skin or less than 5mm to the underlying muscle on the diagnostic scan.
* Any uncontrolled illness or any other medical problem that would preclude surgery.
* The presence of any contraindication for magnetic resonance imaging, e.g. the presence of a heart pacemaker, a metallic foreign body (metal sliver) in the eye, or an aneurysm clip in the brain or severe claustrophobia.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of the HIFU treatment in achieving cancer ablation | 1 month following intervention
  Volume of tumour ablation on histological examination of the surgically excised specimen expressed as a percentage of pretreatment tumour volume on MRI scan.

SECONDARY OUTCOMES:
To evaluate the sensitivity and specificity of post-HIFU MRI in assessing HIFU efficacy when compared with histological evaluation of the resected specimen | 1 month following intervention
  Volume of tumour ablation on histological examination of the surgically excised specimen and volume of tumour ablation on post-treatment MRI expressed as a percentages of pretreatment tumour volume on MRI scan.
Assessment of the safety and toxicity of HIFU ablation | 1 month following intervention
  Using the Common Toxicity Criteria for Adverse Events (CTCAC) Grading Guideline (which scores any occurring adverse events with grades between 1 to 5, where higher grades indicate worse outcomes)
To evaluate patient acceptance of HIFU treatment | 1 month following intervention
  Using 1 to 1 qualitative interviews with participants.

CONTACTS AND LOCATIONS:
Overall Officials: Gurdeep S Mannu, MRCSEd DPhil, Principal Investigator — University of Oxford